CLINICAL TRIAL: NCT02340026
Title: Dynamic Supported Mobility for Infants and Toddlers With Cerebral Palsy
Brief Title: Cerebral Palsy Early Mobility Training
Acronym: iMOVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-011172
Record Dates: First submitted 2015-01-08; First posted 2015-01-16 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Cerebral Palsy
Keywords: Delay in motor skill development
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Therapy (Experimental): The conventional treatment group will receive traditional, therapist-directed pediatric physical therapy. Therapy will focus on early gait training strategies and encouragement of "normal" movement patterns for walking and other age-appropriate movements, with manual guidance or correction of atypical movements from the therapist. This group may use assistive devices, orthoses, and may receive static body weight support for gait training. Therapy activities will be performed in blocks of practice, with the specific activities and level of therapist assistance tailored to each child.
  Interventions: Other: Conventional Therapy
- Dynamic Supported Mobility (Experimental): Children will receive dynamic weight support during all DSM treatment time. The environment will be arranged to encourage active motor exploration, somewhat similar to a play gym for toddlers, to promote the motor variability, engagement, and error experiences that characterize the typical development of upright motor skills and walking. The floor area within 3 feet below either side of the overhead track for a distance of 20 feet (approximately 120 ft2 total) will be defined with colorful thin rubber interlocking mats and arranged with pediatric toys and activities, tailored to the child's interests and to encourage motor skills just beyond his/her current ability. The therapist will minimally assist the child as needed to perform the movements he/she initiates.
  Interventions: Other: Dynamic Supported Mobility

INTERVENTIONS:
Other: Dynamic Supported Mobility — Dynamic weight support; Child-directed; No assistive devices, limited use of orthoses, no treadmill; Encourage high degree of error with reduced physical assistance; Encourage frequent variability in motor tasks (no redirection when moving from one activity to another); Physical therapist expertise is focused on designing a salient and challenging environment for the child's specific interests and ability level to encourage engagement, variability, challenge, and error experience, and on determining the appropriate amount of weight assistance
  Arms: Dynamic Supported Mobility
Other: Conventional Therapy — No or static weight support; Therapist-directed (therapist initiates); Traditional early gait training methods: use of assistive devices/orthoses and may use treadmill; Focus on producing "typical" movement patterns with extensive manual guidance/correction from therapist, prevention of falls; Therapy activities grouped into blocks of practice (i.e. repeated floor to stand practice followed by gait training); Physical therapist expertise is focused on designing and directing the specific practice activities each session, tailored to the individual child
  Arms: Conventional Therapy

SUMMARY:
The purpose of this study is to determine the optimal treatment duration of a novel early mobility training program (dynamic supported mobility, DSM) between 6 to 24 weeks of treatment; and to evaluate the clinical futility of this intervention compared to current rehabilitation practice.

DETAILED DESCRIPTION:
This study is a single-blind, randomized exploratory clinical trial with repeated assessments during a 24-week treatment phase and at three follow-up points over 12 months after treatment to track the developmental trajectory of participants' motor function. Gross motor ability will be compared to published percentile scores of motor function development in cerebral palsy (CP) to determine if the trajectory of predicted motor development is altered, and to outcomes of intensity-matched conventional treatment to determine if continued Phase III investigation is warranted.

ELIGIBILITY:
Inclusion Criteria:

* 12-36 months of age
* Gross motor function below the 10th percentile for age [Bayley Scales of Infant and Toddler Development (BSID), BSID-III, corrected for gestational age, if applicable, under the age of two years].
* Diagnosis of CP or neurological sign associated with CP (i.e. spasticity).
* Ability to initiate pulling to stand at a surface [Score of 1 on gross motor function measure (GMFM) Item 52].
* Cognitive ability to follow one-step commands.

Exclusion Criteria:

* Secondary orthopedic, neuromuscular or cardiovascular condition unrelated to CP.
* General muscle hypotonia, without other neurological signs associated with CP.
* Independent walking ability (Score of 3 on GMFM Item 69 - Walks forward 10 steps).
* At or above the 50th percentile of GMFCS Level I.
* History of surgery or injury to the lower extremities in the past 6 months.

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2020-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Prosser, PT, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Prosser LA, Pierce SR, Skorup JA, Paremski AC, Alcott M, Bochnak M, Ruwaih N, Jawad AF. Motor training for young children with cerebral palsy: A single-blind randomized controlled trial. Dev Med Child Neurol. 2024 Feb;66(2):233-243. doi: 10.1111/dmcn.15729. Epub 2023 Aug 7. PMID 37550991
- [Derived] Pierce SR, Skorup J, Kolobe THA, Smith BA, Prosser LA. Agreement Between the Gross Motor Ability Estimator-2 and the Gross Motor Ability Estimator-3 in Young Children With Cerebral Palsy. Pediatr Phys Ther. 2024 Jan 1;36(1):37-40. doi: 10.1097/PEP.0000000000001065. Epub 2023 Nov 30. PMID 38033276
- [Derived] Prosser LA, Pierce SR, Dillingham TR, Bernbaum JC, Jawad AF. iMOVE: Intensive Mobility training with Variability and Error compared to conventional rehabilitation for young children with cerebral palsy: the protocol for a single blind randomized controlled trial. BMC Pediatr. 2018 Oct 16;18(1):329. doi: 10.1186/s12887-018-1303-8. PMID 30326883

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from January 2015 through January 2019. The primary sources of recruitment were the Cerebral Palsy, outpatient physical therapy and Neonatal Follow-up programs at our institution.
Pre-assignment Details: Full baseline assessment not completed (n=1)
Groups:
- Dynamic Supported Mobility (DSM): Children will receive dynamic weight support during all Dynamic Supported Mobility (DSM) treatment time. The environment will be arranged to encourage active motor exploration, somewhat similar to a play gym for toddlers, to promote the motor variability, engagement, and error experiences that characterize the typical development of upright motor skills and walking. The floor area within 3 feet below either side of the overhead track for a distance of 20 feet (approximately 120 ft2 total) will be defined with colorful thin rubber interlocking mats and arranged with pediatric toys and activities, tailored to the child's interests and to encourage motor skills just beyond his/her current ability. The therapist will minimally assist the child as needed to perform the movements he/she initiates.
  Dynamic Supported Mobility: Dynamic weight support; Child-directed; No assistive devices, limited use of orthoses, no treadmill; Encourage high degree of error with reduced physical assistance; Encourage frequent variability in motor tasks (no redirection when moving from one activity to another); Physical therapist expertise is focused on designing a salient and challenging environment for the child's specific interests and ability level to encourage engagement, variability, challenge, and error experience, and on determining the appropriate amount of weight assistance
Period: Treatment Phase
Arm/Group | Conventional Therapy | Dynamic Supported Mobility (DSM)
Started | 21 | 20
Completed | 19 | 18
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2
Period: Follow-up Phase
Arm/Group | Conventional Therapy | Dynamic Supported Mobility (DSM)
Started | 19 | 18
Completed | 18 | 18
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Therapy | Dynamic Supported Mobility | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21 | 20 | 41
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 23.2 (7.2) | 20.4 (5.1) | 21.8 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 11 | 12 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 19 | 17 | 36
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 7 | 10
  White | 15 | 12 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 20 | 41
Gross Motor Function Classification System (GMFCS) [Count of Participants; unit: Participants] — GMFCS level descriptions (once school age):
  LEVEL I Walks without Limitations LEVEL II Walks with Limitations LEVEL Ill Walks Using a Hand-Held Mobility Device LEVEL IV Self-Mobility with Limitations; May Use Powered Mobility LEVEL V Transported in a Manual Wheelchair
  Participants
    I | 3 | 2 | 5
    II | 9 | 8 | 17
    III | 5 | 5 | 10
    IV | 4 | 5 | 9
    V | 0 | 0 | 0
Anatomical typography [Count of Participants; unit: Participants]
  Monoplegia | 0 | 1 | 1
  Hemiplegia | 5 | 3 | 8
  Diplegia | 10 | 8 | 18
  Triplegia | 1 | 2 | 3
  Quadriplegia | 4 | 6 | 10
  Unknown | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Gross Motor Function Measure (GMFM-66) During Treatment Phase
Description: Computation of the GMFM-66 score involves statistical weighting of the raw item scores for difficulty. This score will also be used with the patient's age to determine Gross Motor Function Classification System (GMFCS) percentile rank. Scores range from 0 (no volitional movement) to 100 (gross motor function of an average 5 year old). Higher scores reflect better outcomes.
Time Frame: Baseline and 12 weeks
Population: Participants with completed baseline and 12 week assessments
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conventional Therapy | Dynamic Supported Mobility
Number analyzed (Participants) | 19 | 18
units on a scale | 2.2 (3.2) | 3.5 (2.6)

2. Secondary Outcome: Change in Postural Control
Description: Early Clinical Assessment of Balance - a clinical test of balance and postural control developed for administration with young children. The minimum score is 0. The maximum score is 100. Higher scores reflect better postural control.
Time Frame: Baseline and 12 weeks
Population: All participants with baseline and 12 week scores
Measure: Mean (Standard Deviation); unit: ECAB score units
Arm/Group | Conventional Therapy | Dynamic Supported Mobility
Number analyzed (Participants) | 19 | 18
ECAB score units | 2.7 (4.7) | 4.3 (5.9)

3. Secondary Outcome: Change in Physical Activity
Description: A wireless activity monitor will be provided to the caregiver, who will be instructed on use of the monitor at home, with a goal of recording 5 total hours of the child's free play in the following week. Amount and magnitude of physical activity will be calculated from the acceleration time series using signal processing software.
Time Frame: Weeks 0 and 12
Population: All participants with evaluable data from using the wearable sensors at home at Times 0 and 12 weeks.
Measure: Mean (Standard Deviation); unit: change in percent active time
Arm/Group | Conventional Therapy | Dynamic Supported Mobility (DSM)
Number analyzed (Participants) | 9 | 7
change in percent active time | 1.4 (8.9) | -2.6 (11.5)

4. Secondary Outcome: Change in Caregiver Satisfaction
Description: Using the Canadian Occupational Performance Measure, one caregiver of each participant will rate their child's performance on the caregiver's self-identified goals, and then rate their own (caregiver's) satisfaction with the child's performance. Satisfaction is rated on a scale of 1-10, with higher ratings reflecting greater parent satisfaction.
Time Frame: Baseline and 12 weeks
Population: All participants with baseline and 12 week scores
Measure: Mean (Standard Deviation); unit: COPM score units
Arm/Group | Conventional Therapy | Dynamic Supported Mobility
Number analyzed (Participants) | 19 | 18
COPM score units | 1.5 (2.7) | 2.5 (2.8)

5. Secondary Outcome: Change in Child Engagement in Daily Life
Description: One caregiver of each participant will complete the Child Engagement in Daily Life Measure to obtain a measure of the child's participation in play in daily life. Scaled scores range from 0-100. Higher scores reflect greater engagement in daily life.
Time Frame: Baseline and 12 weeks
Population: All participants with baseline and 12 week scores
Measure: Mean (Standard Deviation); unit: CEDL scaled score units
Arm/Group | Conventional Therapy | Dynamic Supported Mobility
Number analyzed (Participants) | 18 | 18
CEDL scaled score units | 0.96 (7.1) | 3.8 (6.1)

ADVERSE EVENTS:
Time Frame: Enrollment to study completion (up to 18 months)
Arm/Group | Conventional Therapy | Dynamic Supported Mobility
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 3/21 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Therapy (N=21) | Dynamic Supported Mobility (N=20)
Fall in a toddler (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) — Developmentally-appropriate falls in our toddler age cohorts. The child needed a 1-5 minute break after the fall, then resumed study procedures as planned. Three falls occurred during a treatment session, one occurred during an assessment session.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-23): https://cdn.clinicaltrials.gov/large-docs/26/NCT02340026/Prot_SAP_000.pdf